CLINICAL TRIAL: NCT06057376
Title: Clinical Comparison of the Impact of Two Dietary Interventions on Abdominal Pain and Intestinal Microbiome Caused by Simple Carbohydrate Intolerance.
Brief Title: Impact of Two Dietary Interventions on Simple Carbohydrate Intolerance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Oregon (Other); Oregon State University (Other)
Responsible Party: Principal Investigator, Anna Hunter, MD, MCR, MD, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB No.24928
Record Dates: First submitted 2023-09-15; First posted 2023-09-28 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Carbohydrate Intolerance
MeSH Terms: conditions — Glucose-Galactose Malabsorption | interventions — lipoic acid synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low FODMAP group (Other): Participants randomized to this group will be instructed based on published low-FODMAP diet guidelines and provided with sample meal plans to aid in compliance. Each participant will be randomized to low-FODMAP diet group (LFD) for 3 weeks.
  Interventions: Other: Low-FODMAP diet group (LFD)
- Low Added Sugar group (Other): Each participant will be randomized to either the low-FODMAP diet group (LFD) or the low added sugar diet group (LAS) for 3 weeks. Each participant will be randomized to the low added sugar diet group (LAS) for 3 weeks.
  Interventions: Other: Low Sugar diet group (LAS)

INTERVENTIONS:
Other: Low-FODMAP diet group (LFD) — Each participant will be following a low-FODMAP diet group for 3 weeks, followed by 3 week break prior to second diet intervention.
  Arms: Low FODMAP group
Other: Low Sugar diet group (LAS) — Each participant will be following a low added sugar diet group for 3 weeks, after 3 week break.
  Arms: Low Added Sugar group

SUMMARY:
In this project we want to assess impact of dietary fructose as a simple sugar intolerance on abdominal pain and compare a low FODMAP diet versus an added sugar elimination diet effectiveness on symptoms but also impact on microbiome and its metabolome.

DETAILED DESCRIPTION:
This is a prospective cross over study. Participants who meet the study entry criterion, will be randomized to a specific dietary intervention: low FODMAP for a 3-week period or Limited Added Sugar for 3 weeks. After the initial study phase, participants will enter a 3 week break followed by a crossover to the other diet phase.

Each participant will be randomized to either the low-FODMAP diet group (LFD) or the low added sugar diet group (LAS) for 3 weeks. All participants will be assigned to a nutrition intervention consisting of 2 one-hour counseling sessions (pre and post diet initiation) plus one 30 min telephone session at week 1 and 2 of the intervention for both diet groups. Macronutrients will not be restricted and both study diets will be ad libitum. Diet interventions will include administration of a 24 hour food recall and completion of the Comprehensive Nutrition Assessment Questionnaire in addition to comprehensive education of the assigned diet.

Investigators will collect stool samples prior to intervention and post each diet intervention to assess initial microbiome composition as well as post intervention changes. Symptom data will be collected via an online survey link consisting of abdominal pain related questionnaires. Measures for child and parent will be requested at the time enrollment of the study and at the end of each diet phase.

Animal studies indicate microbiome adjustment to an increase in dietary carbohydrate pool. It is difficult to capture this change in humans as the microbiome shift may not be evident by actual change in certain strains but by genomic adjustment. Investigators propose a metagenomic approach in combination with metabolomics to identify microbiome end products present as a result of changes in dietary carbohydrate intake by dietary elimination.

Investigators will characterize shifts in metagenomic composition in response to dietary shifts using multivariate methods and linear mixed effects models. To address our hypothesis that FODMAP and low added sugar diets will affect microbial gene content in similar ways, investigators will compare metagenomic shifts relative to a baseline diet using multivariate models that control for subject, age, sex, diet order and potential confounding factors in PerMANOVA and distance-based redundancy analyses. Investigators will have 95% power to detect medium shifts in metabolic profiles among dietary groups (Cohen's D = 0.520). Investigators will use mixed effect linear models to measure enrichment for specific metabolic pathways and diet-driven shifts in specific metabolites over time while controlling for subject, age, sex, diet order, symptoms and potential confounding factors. In these repeated measures design, we will have 95% power to detect a small to medium effect of diet on a given metabolite (Cohen's D = 0.371). The Benhamini-Hochberg procedure will be applied to decrease the false discovery rate when running multiple tests (Yoav et al) It is also of interest to analyze how microbial gene content and metabolic profiles covary. Investigators will apply qualitative genetic methods of covariance matrix estimation to determine how metabolite profiles can be predicted by metagenomic content.

ELIGIBILITY:
Inclusion Criteria:

* Age: 5- 18-year-old
* BMI: within normal range for age
* Positive fructose breath test performed as part of diagnostic work up for abdominal pain
* Willingness to consume low FODMAP and Limited Added sugar diet trial and collect required samples

Exclusion Criteria:

* Age: not within range
* BMI: not within range
* Negative fructose breath test
* Any known or suspected intestinal disorder including but not limited to IBD, IBS, celiac disease, Crohn's Disease, food sensitivities, food allergies, significant by-choice food restrictions
* Hormonal disorders
* Use of chronic medications including contraceptives (both oral and subcutaneous), non-hormone secreting IUD- accepted
* Use of oral or IV antibiotics in the last three months
* Daily probiotic use (pill form)
* Daily multi-vitamin except vitamin D supplements

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Abdominal Pain | 63 days
  Diet impact on abdominal pain as assessed by a questionnaire before and after each diet intervention
Effect of each diet on microbiome and metabolome | 63 days
  Impact of each diet intervention on microbiome and metabolome will be assessed utilizing a stool sample collected prior to and after diet completion

CONTACTS AND LOCATIONS:
Overall Officials: Anna Hunter, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Springfield, Oregon, United States